CLINICAL TRIAL: NCT07070427
Title: The Effect of Cognitive-Based Balance Exercises on the Shooting Performance of Archers
Brief Title: Cognitive-Based Balance Exercises on the Shooting Performance of Archers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1301MA-001
Record Dates: First submitted 2025-05-09; First posted 2025-07-17 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Archery; Cognitive Performance; Balance Training
Keywords: shooting performance; static balance; dynamic balance; cognitive
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventions (Experimental): Participants performed balance exercises twice a week for 12 weeks using the BOSU balance ball. The exercises included static and dynamic balance tasks. Additionally, during dual-task training, cognitive tasks such as counting backwards, naming months and days of the week in reverse order, and identifying numerical differences were incorporated alongside balance exercises. Archery performance was assessed by shooting 5 sets of 3 arrows at a target from a distance of 18 meters, both before and after the intervention.
  Interventions: Other: Exercise
- Control (Experimental): Participants performed the same balance exercises twice a week for 12 weeks using the BOSU balance ball, focusing on static and dynamic balance tasks without additional cognitive tasks. Archery performance was evaluated in the same manner as the experimental group, shooting 5 sets of 3 arrows at a target 18 meters away, before and after the training period.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Cognitive-based balance exercises.

SUMMARY:
The aim of this treatment study is to determine the effects of cognitive-based balance exercises on archers' shooting performance. The study focuses on archers and examines the effects of cognitive-based dynamic and static balance exercises on shooting accuracy.

In this context, the main questions that the study aims to answer are as follows:

* Cognitive-based balance exercises applied to archers have no effect on shooting performance.
* Cognitive-based balance exercises applied to archers have an effect on shooting performance.

The researchers will evaluate the effects of the interventions on shooting performance by comparing the performance differences between archers who apply cognitive-based balance exercises and archers who only do balance exercises.

Participants:

* The control group will apply various balance exercises during the 12-week training period. The study group will apply cognitive-based balance exercises.
* They will be subjected to performance tests that evaluate static balance, dynamic balance and shooting accuracy.

DETAILED DESCRIPTION:
This study investigates the effects of cognitive-based balance training on archery performance by targeting not only shooting accuracy, but also neuromuscular and sensorimotor parameters such as shoulder joint position sense and bilateral upper extremity force symmetry. While conventional balance exercises primarily focus on postural control and neuromuscular coordination, cognitive-based balance training integrates executive functions-such as attention, working memory, and decision-making-into postural tasks, aiming to enhance cognitive-motor coupling and sensorimotor integration.

The training program is designed to include both static and dynamic balance activities combined with cognitively demanding tasks, such as dual-tasking, response inhibition, and visuospatial challenges. Progression and supervision are employed to maintain intervention fidelity throughout the 12-week period. Archery performance will be assessed pre- and post-intervention using standardized shooting accuracy protocols.

To further investigate potential mechanisms underlying performance changes, two additional neuromuscular variables will be evaluated. Shoulder proprioception will be assessed using a digital clinometer through passive position-reproduction tests in multiple planes of motion (e.g., flexion, abduction, and internal/external rotation at specific angles). This will help determine whether improvements in sensorimotor function accompany changes in performance. Bilateral force symmetry will be assessed using a digital hand dynamometer by comparing maximal isometric grip strength in unilateral and bilateral conditions. The resulting bilateral deficit values will offer insight into interlimb coordination and neural efficiency.

By combining cognitive, postural, and upper extremity neuromuscular assessments, this study aims to provide a comprehensive understanding of how cognitively enriched balance interventions may influence both central and peripheral components of athletic performance in archery. The findings are expected to contribute to the growing literature on cognitive-motor integration in precision sports and inform future training paradigms in disciplines that demand both motor accuracy and cognitive control.

ELIGIBILITY:
Inclusion Criteria:

* Being a licensed archery athlete,
* Having been practicing archery for at least 2 years,
* Participating in a training program at least 2 days a week,
* Using a compound bow,
* Being between the ages of 18-45.

Exclusion Criteria:

* Having any diagnosed lung, cardiovascular, neurological, systemic and orthopedic disease,
* Receiving conservative or surgical treatment after trauma in the upper and lower extremities,
* Having had a musculoskeletal injury within the last year,
* Using corticosteroids or any other medication,
* Having a psychological dysfunction.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-09-23 (Estimated)

PRIMARY OUTCOMES:
Static and Dynamic Balance Exercise Training | 5-6 minutes
  Duration and Type of Static and Dynamic Balance Exercises Using BOSU Balance Ball (minutes) Static and dynamic balance exercises were performed using the BOSU balance ball to enhance proprioception. Exercises included maintaining balance for 30 seconds with eyes open or closed in various positions: static standing with one foot crossed over the other, single-leg standing, gliding stance, double-foot tiptoe rise, and multi-directional reaching while balancing on one foot (right and left) on the BOSU ball. This training protocol was applied to both the control and experimental groups.
Evaluation of Dynamic Balance: | 5 minutes
  Y-Balance Test Reach Distance (centimeter) Description: Dynamic balance was assessed by measuring the maximum reach distance (in centimeters) during the Y-Balance Test at baseline and after 12 weeks of training.
Evaluation of Static Balance | 5 minutes
  Standing Stork Test Duration (seconds) Description: Static balance was evaluated by measuring the duration (in seconds) participants were able to maintain a one-legged stance during the Standing Stork Test at baseline and post-intervention.
Dual Task Training | 10 minutes
  Performance on Cognitive Tasks During Balance Exercises (e.g., counting backwards, reverse recitation) Participants in the study group performed cognitive tasks simultaneously with balance exercises. Tasks included counting backwards by 7 while standing statically, reciting months in reverse while standing on one leg, stating the preceding number when given a number between 1 and 100 during tandem stance, listing days of the week in reverse while standing on tiptoe, and naming 5 words starting with a given letter while reaching in multiple directions on one leg.
Evaluation of Shooting Performance | 5 minutes
  Total Archery Performance Score (points scored in 5 sets of 3 arrows at 18 meters) Archery performance was measured by the total points scored when participants shot 5 sets of 3 arrows at a target 18 meters away. Assessments were conducted at baseline and after 12 weeks of balance training.ce training.
Evaulation of Joint Position Sense | 3 minutes
  Mean Angular Error in Shoulder Joint Position Reproduction Test (degrees) Shoulder joint position sense was assessed using a passive position-reproduction test with a digital clinometer. Participants were passively positioned at predetermined angles and asked to actively replicate the position with eyes closed. Angular deviations (in degrees) from the target position were recorded. Measurements were taken for shoulder flexion, abduction (standing), and external/internal rotation at 90° abduction (supine). The mean error was calculated based on three repetitions for each movement. Tests were performed by two independent assessors on the same day to ensure reliability.
Evaluation of Bilateral Deficit | 2 minutes
  Percentage Bilateral Deficit in Maximal Isometric Grip Strength (%)
  Bilateral deficit of upper extremity muscle strength was assessed using a digital hand dynamometer. Participants performed three maximal isometric grip trials with each hand separately and three simultaneous bilateral maximal isometric grip trials. The bilateral deficit (%) was calculated using the formula:
  Bilateral Deficit (%) = ((Right Hand + Left Hand) - Bilateral Force) / (Right Hand + Left Hand) × 100.
  Positive values indicate bilateral deficit; negative values indicate bilateral facilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Sema ÖZDEN ACARÖZ, Msc, Principal Investigator — Cyprus International University
Locations (1):
- Cyprus International University, Mersin, Lefkosa, Turkey (Türkiye)

REFERENCES:
- See also: On-target trajectories and the final pull in archery — https://www.researchgate.net/publication/233046298_On-target_trajectories_and_the_final_pull_in_archery
- See also: Dynamic stretching is effective as static stretching at increasing flexibility — https://www.researchgate.net/publication/321890007_Dynamic_stretching_is_effective_as_static_stretching_at_increasing_flexibility
- See also: Postural Sway Distinguishes Shooting Accuracy among Skilled Recurve Archers — https://doi.org/10.15282/mohe.v1i0.5
- See also: Anthropometric And Physical Fitness Components Comparison between High- And Low-Performance Archers — https://www.researchgate.net/publication/348825411_Anthropometric_And_Physical_Fitness_Components_Comparison_between_High-_And_Low-Performance_Archers
- See also: Sensorimotor System Measurement Techniques — https://www.researchgate.net/publication/7219971_Sensorimotor_System_Measurement_Techniques
- See also: Comparison of Modular Control of Trunk Muscle by Japanese Archery Competitive Level: A Pilot Study — https://www.jstage.jst.go.jp/article/ijshs/15/0/15_201714/_article
- See also: Biomechanics Measurements in Archery — https://www.researchgate.net/publication/269914195_Biomechanics_Measurements_in_Archery
- See also: Proprioception and balance training can improve amateur soccer players' technical skills — https://www.researchgate.net/publication/286020065_Proprioception_and_balance_training_can_improve_amateur_soccer_players'_technical_skills
- See also: Correlation among proprioception, muscle strength, and balance — https://pubmed.ncbi.nlm.nih.gov/28174475/
- See also: https://pubmed.ncbi.nlm.nih.gov/29097947/ — https://pubmed.ncbi.nlm.nih.gov/29097947/
- See also: Age-related shift in neural complexity related to task performance and physical activity — https://pubmed.ncbi.nlm.nih.gov/25244121/
- See also: The Effects of Physical Exercise and Cognitive Training on Memory and Neurotrophic Factors — https://pubmed.ncbi.nlm.nih.gov/28699808/
- See also: Balance Expertise Is Associated with Superior Spatial Perspective-Taking Skills — https://pmc.ncbi.nlm.nih.gov/articles/PMC8615958/
- See also: Training effects on motor-cognitive dual-task performance in older adults — https://eurapa.biomedcentral.com/articles/10.1007/s11556-013-0122-z
- See also: Injury History, Sex, and Performance on the Functional Movement Screen and Y Balance Test — https://pmc.ncbi.nlm.nih.gov/articles/PMC4495982/
- See also: The Relationship Between Maximum Unilateral Squat Strength and Balance in Young Adult Men and Women — https://pmc.ncbi.nlm.nih.gov/articles/PMC3827570/
- See also: Target Archery | World Archery. https://worldarchery.org/TargetArchery#INDOOR. Accessed May 11, 2020. — https://www.worldarchery.sport/archeryplus?gad_source=1&gclid=CjwKCAjwp8--BhBREiwAj7og16_kBDjZy14zhJMuyLzGY3VGb8uxVLUOLgEUGiwitE7ap3V59iPqgRoC3AQQAvD_BwE